CLINICAL TRIAL: NCT03373331
Title: Treating Emotional Processing Impairments in Individuals With TBI: A Randomized Controlled Trial
Brief Title: Treating Emotional Processing Impairments in Individuals With TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Commission on Brain Injury Research (Other)
Responsible Party: Principal Investigator, Helen Genova, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-875-15
Record Dates: First submitted 2017-12-08; First posted 2017-12-14 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Brain Injury
Keywords: Emotional Processing; Cognition; Traumatic Brain Injury; Intervention
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Participants in the experimental group will receive emotional processing training exercises administered on a laptop computer. They will undergo 12 sessions of 45-60 minutes each (twice a week for 6 weeks).
  Interventions: Behavioral: Emotional Processing Training
- Control Group (Placebo Comparator): Participants in the control group will meet with the examiner the same frequency and for the same duration as those in the experimental group.
  They will receive placebo control exercises administered on a laptop computer.
  .
  Interventions: Behavioral: Placebo Control Exercises

INTERVENTIONS:
Behavioral: Emotional Processing Training — Participants in the experimental group will receive computerized exercises administered on a laptop computer. They will undergo 12 sessions of 45-60 minutes each (twice a week for 6 weeks).
  Arms: Experimental Group
Behavioral: Placebo Control Exercises — Participants in the control group will receive computerized control exercises administered on a laptop computer. They will undergo 12 sessions of 45-60 minutes each (twice a week for 6 weeks).
  Arms: Control Group

SUMMARY:
The current project will examine the impact of an emotional processing intervention on emotional processing abilities in a sample of 50 persons with moderate to severe TBI. Outcome will be assessed across 3 domains. We will document changes resulting from treatment: (1) in emotional processing tasks (2) in other areas of function including QOL, social functioning, mood and cognition that are also likely to be impacted (3) in brain structure and function. The examination of efficacy in the above three areas will further our knowledge of emotional processing deficits in TBI and more importantly, identify an effective means of treating such deficits.

DETAILED DESCRIPTION:
Emotional processing deficits have a significant negative impact on the lives of persons with TBI. There is emerging research indicating that, in addition to cognitive and behavioral impairments, social and emotional difficulties following TBI are common and are related to significant problems in social relationships, poor social participation, impaired empathy, and a high degree of caregiver stress. Emotional processing is a critical component of social cognition, including the abilities to both identify and discriminate basic universal emotions. The stability of emotional processing deficits following TBI indicates that these impairments likely impact individuals with TBI consistently across the lifespan, and do not appear to resolve with time.

The goals of the trial are to (a) Evaluate the effectiveness of an emotional processing intervention to improve performance on tests of emotional processing in individuals with TBI, (b) Evaluate the improvement of secondary outcomes of psychological, cognitive, and functional abilities following the emotional processing intervention in individuals with TBI, (c) To examine differences in brain activation patterns during emotional processing following treatment in individuals with TBI, BOLD activation in the experimental group will be compared to BOLD patterns of the control group during performance of the QFDT, a facial affect recognition task.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Traumatic Brain Injury (TBI)
* can read and speak English fluently

Exclusion Criteria:

* prior stroke or neurological disease.
* history of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder, Schizophrenia, Epilepsy, Bipolar Disorder
* significant alcohol or drug abuse history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Facial Expression Identification Task (FEIT) | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  The FEIT assesses one's ability to correctly identify and discriminate emotions from faces.

SECONDARY OUTCOMES:
Emotion Regulation Questionnaire (ERQ) | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  The ERQ is a self-report measure of the use of 2 emotional regulation strategies: cognitive reappraisal and expressive suppression.
Satisfaction with Life Scale (SWLS) | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  The SWLS is a self-report measure of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Genova, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States